CLINICAL TRIAL: NCT03073369
Title: Targeting the Interactions Between Disordered Iron Homeostasis and Mineral Metabolism in Chronic Kidney Disease (Aim 1)
Brief Title: Effect of Ergocalciferol on Iron Metabolism in Individuals With Chronic Kidney Disease
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study didn't materialize for various reasons.
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Bhupesh Panwar, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: F170216006
Record Dates: First submitted 2017-02-28; First posted 2017-03-08 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: CKD; Chronic Kidney Diseases; Hepcidin; Ergocalciferol; Vitamin D; Iron-deficiency; Anemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia, Iron-Deficiency; Anemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oral Ergocalciferol (Active Comparator): Oral Ergocalciferol 50000 IU once daily for 6 weeks
  Interventions: Drug: Ergocalciferol 50000 UNT
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ergocalciferol 50000 UNT — Oral Ergocalciferol 50000 IU once daily for 6 weeks
  Arms: Oral Ergocalciferol
Drug: Placebo — Oral Placebo - one capsule once daily for 6 weeks
  Arms: Placebo

SUMMARY:
The purpose of the study is to learn more about how treatment with vitamin D can affect iron metabolism and blood levels of hepcidin (hormone controlling iron levels) in people with chronic kidney disease (CKD).

Iron is an essential mineral which is a major component of proteins that carry oxygen in the blood. Problems with iron metabolism can lead to low blood levels (anemia), which can commonly happen in people with CKD.

New research over the last decade has uncovered a new hormone called 'hepcidin', which is made in the liver and released into the blood. Hepcidin controls how much iron is in the blood by preventing the absorption of iron from food. Blood levels of hepcidin C are found to be high in people with CKD, and a recent small study in people with normal kidney function showed that treatment with vitamin D decreased hepcidin levels.

In this study, investigators would like to examine the effects of vitamin D (Ergocalciferol) on iron metabolism and blood levels of hepcidin in individuals with CKD.

ELIGIBILITY:
Inclusion Criteria:

* Participants 19 years or older with mild to moderate CKD (eGFR 15 - 59 ml/min/1.73 m2) by the CKD-EPI formula, with vitamin D deficiency (25(OH)D < 30 ng/ml), and with absolute iron deficiency (TSAT < 20 and Ferritin <100) or iron restriction (TSAT < 20 and Ferritin > 100).

Exclusion Criteria:

* Active vitamin D analog therapy or history of recent (< 3 months) use.
* Nutritional vitamin D (cholecalciferol or ergocalciferol) therapy in dosages greater than 2000 IU/day.
* Subjects receiving erythropoiesis stimulating agents or intravenous iron therapy.
* Oral iron therapy started within the last 3 months.
* Hb < 8.0 g/dL for males and Hb <7.0 g/dL for females.
* Pregnancy or lactation.
* Serum calcium > 10.0 mg/dL or phosphorus > 4.5 mg/dL.
* Subjects with acute kidney injury or rapidly declining GFR.
* Subjects on hemodialysis, peritoneal dialysis, or having a functioning renal transplant.
* Focus of active inflammation such as acute gout, rheumatoid arthritis or active infection determined clinically.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in serum hepcidin levels | At Day 0, Day 3, 1 week, 4 weeks and 6 weeks
  Difference in change in serum hepcidin levels (ng/ml) over time between the two groups

SECONDARY OUTCOMES:
Change in serum hemoglobin level | At Day 0, Day 3, 1 week, 4 weeks and 6 weeks
  Difference in change in serum hemoglobin levels (g/dL) over time between the two groups
Change in serum ferritin level | At Day 0, Day 3, 1 week, 4 weeks and 6 weeks
  Difference in change in serum ferritin levels (ng/ml) over time between the two groups
Change in percent transferrin saturation | At Day 0, Day 3, 1 week, 4 weeks and 6 weeks
  Difference in change in percent transferrin saturation (%) over time between the two groups
Change in serum iron level | At Day 0, Day 3, 1 week, 4 weeks and 6 weeks
  Difference in change in serum iron levels (mcg/dL) over time between the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No